CLINICAL TRIAL: NCT05334108
Title: A Phase 1, Open-Label, Fixed Sequence, Drug-Drug Interaction Study to Evaluate the Effects of Repeat Titrated Doses of Ecopipam on the Pharmacokinetics of Multiple Substrates for Drug Metabolism and Transport in Healthy Subjects
Brief Title: Drug-Drug Interaction Study to Evaluate the Effects of Ecopipam on the Pharmacokinetics of Multiple Substrates for Drug Metabolism and Transport
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: ICON Early Phase Services (Unknown); Nuventra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EBS-101-HV-104
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Drug Interaction
MeSH Terms: interventions — ecopipam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): ecopipam HCl oral tablets of 12.5, 50, 75, and 100 mg daily for up to 20 days
  Cohort 1 Probe Substrate Cocktail given on 2 separate days:
  * midazolam: 1 µg infused IV
  * caffeine: 200 mg oral tablet
  * omeprazole: two 20 mg oral tablets
  * dextromethorphan: 1.6mL (containing ~10 mg) oral solution
  Interventions: Drug: Ecopipam; Combination Product: Cohort 1 Probe Substrate Cocktail
- Cohort 2 (Other): ecopipam HCl oral tablets of 12.5, 50, 75, and 100 mg daily for up to 20 days
  Cohort 2 Probe Substrate given on 2 separate days:
  - bupropion: 100mg oral tablet
  Interventions: Drug: Ecopipam; Drug: Cohort 2 Probe Substrate
- Cohort 3 (Other): ecopipam HCl oral tablets of 12.5, 50, 75, and 100 mg daily for up to 20 days
  Cohort 3 Probe Substrate Cocktail given on 3 separate days:
  * midazolam: 10 µg/mL given as 1mL oral solution.
  * dabigatran: 375 µg/mL and pitavastatin: 10 µg/mL given as 1mL oral solution
  * rosuvastatin: 25 µg/mL and atorvastatin: 50 µg/mL given as 2mL oral solution
  Interventions: Drug: Ecopipam; Combination Product: Cohort 3 Probe Substrate Cocktail

INTERVENTIONS:
Drug: Ecopipam — ecopipam HCl ~2mg/kg/day
Combination Product: Cohort 1 Probe Substrate Cocktail — dextromethorphan, caffeine, omeprazole, and midazolam
  Arms: Cohort 1
Drug: Cohort 2 Probe Substrate — bupropion
  Arms: Cohort 2
Combination Product: Cohort 3 Probe Substrate Cocktail — dabigatran, pitavastatin, rosuvastatin, atorvastatin, midazolam
  Arms: Cohort 3

SUMMARY:
This is a single center, open-label, fixed sequence Phase 1, drug-drug interaction (DDI) study in healthy subjects.

DETAILED DESCRIPTION:
Following a Screening period, eligible subjects will be enrolled sequentially to one of three cohorts to receive a single dose of probe substrate(s), followed by repeated titrated doses of ecopipam twice daily (BID) (with subjects in Cohort 3 also receiving a single dose of ecopipam and probe substrates on Day 4 prior to titration). After steady-state ecopipam dosing is reached, ecopipam will be co-administered with a single dose of probe substrate(s) (with continuation of ecopipam BID (every 12 h) dosing during the blood sampling period for the respective probe substrates), followed by an ecopipam tapering period and clinic discharge assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or female subjects of non-childbearing potential
* ≥18 and <55 years of age at the time of consent
* BMI >18.5 and <30 kg/m2 and a weight of ≥50 kg for males or ≥45 kg for females
* Subjects must be healthy, as determined by the Investigator, based on medical history, physical examination, ECG, and standard panel of blood and laboratory tests at Screening.
* Sexually active males must use a double barrier method of contraception during the study and for at least 90 days after the last dose of study drug
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration

Exclusion Criteria:

* Personal or family History of significant medical illness
* Clinically significant abnormalities on screening tests/exams
* History of or significant risk of committing suicide
* Donation of plasma within 7 days prior to dosing
* Donation or significant loss of blood within 30 days prior to the first dosing
* Major surgery within 3 months or minor surgery within 1 month prior to admission
* Use of prohibited prescription, over-the-counter medications or natural health products
* Alcohol-based products 24 hours prior to admission
* Female subjects who are currently pregnant or lactating
* Positive pregnancy test
* Use of tobacco or nicotine products within 3 months prior to Screening
* Significant alcohol consumption
* History of drug abuse within the previous 2 years, or a positive drug screen
* History of allergy to study medications
* Undergoing abrupt discontinuation of alcohol or sedatives
* Not suitable for study in the opinion of the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Cmax of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of dabigatran in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of dabigatran in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of rosuvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of rosuvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of dabigatran in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of dabigatran in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of rosuvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of rosuvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of dabigatran in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of dabigatran in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of rosuvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of rosuvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of dabigatran in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of dabigatran in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of rosuvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of rosuvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-24 of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis

SECONDARY OUTCOMES:
Cmax of bupropion (and its 4-hydroxybupropion metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of bupropion (and its 4-hydroxybupropion metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax omeprazole (and its 5'-hydroxy omeprazole metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax omeprazole (and its 5'-hydroxy omeprazole metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of bupropion (and its 4-hydroxybupropion metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of bupropion (and its 4-hydroxybupropion metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of bupropion (and its 4-hydroxybupropion metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of bupropion (and its 4-hydroxybupropion metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dextromethorphan in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dextromethorphan in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL for IV midazolam in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL for IV midazolam in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for oral midazolam in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for oral midazolam in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dabigatran in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dabigatran in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for pitavastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for pitavastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for rosuvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for rosuvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for atorvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for atorvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for bupropion in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for bupropion in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for caffeine in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for caffeine in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for omeprazole in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for omeprazole in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dextromethorphan in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dextromethorphan in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V for IV midazolam in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V for IV midazolam in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for oral midazolam in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for oral midazolam in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dabigatran in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dabigatran in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for pitavastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for pitavastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for rosuvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for rosuvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for bupropion in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for bupropion in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for atorvastatin in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for atorvastatin in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for caffeine in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for caffeine in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for omeprazole in the presence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for omeprazole in the absence of ecopipam | Up to Day 22
  Up to 46 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Total concentration of bilirubin in the presence of ecopipam | Up to Day 18
  Bilirubin sampling will occur on Day 1 and Day 18
Total concentration of bilirubin in the absence of ecopipam | Up to Day 18
  Bilirubin sampling will occur on Day 1 and Day 18
Unconjugated concentration of bilirubin in the presence of ecopipam | Up to Day 18
  Bilirubin sampling will occur on Day 1 and Day 18
Unconjugated concentration of bilirubin in the absence of ecopipam | Up to Day 18
  Bilirubin sampling will occur on Day 1 and Day 18
Conjugated concentration of bilirubin in the presence of ecopipam | Up to Day 18
  Bilirubin sampling will occur on Day 1 and Day 18
Conjugated concentration of bilirubin in the absence of ecopipam | Up to Day 18
  Bilirubin sampling will occur on Day 1 and Day 18
Average of the 6-hour plasma dextromethorphan: dextrorphan ratio in the presence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 8-hour plasma dextromethorphan: dextrorphan ratio in the presence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 12-hour plasma dextromethorphan: dextrorphan ratio in the presence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 6-hour plasma dextromethorphan: dextrorphan ratio in the absence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 8-hour plasma dextromethorphan: dextrorphan ratio in the absence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 12-hour plasma dextromethorphan: dextrorphan ratio in the absence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 6-hour plasma caffeine: paraxanthine metabolite ratio in the presence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 8-hour plasma caffeine: paraxanthine metabolite ratio in the presence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 12-hour plasma caffeine: paraxanthine metabolite ratio in the presence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 6-hour plasma caffeine: paraxanthine metabolite ratio in the absence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 8-hour plasma caffeine: paraxanthine metabolite ratio in the absence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Average of the 12-hour plasma caffeine: paraxanthine metabolite ratio in the absence of ecopipam | Up to Day 14
  6 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Safety and tolerability as demonstrated by the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) | Up to Day 63
  Score from 0-5 where 0 is no response and 5 is responds readily. MOAA/S measures will be recorded at the indicated timepoints
Safety and tolerability as demonstrated by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Day 63
  Safety and tolerability measures will be recorded at the indicated timepoints
Number of participants requiring concomitant medications | Up to Day 63
  Participants will be continuously monitored for the use of concomitant medications
AEs with relatedness associated with dextromethorphan | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with IV midazolam | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with oral midazolam | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with dabigatran | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with pitavastatin | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with rosuvastatin | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with atorvastatin | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with bupropion | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with caffeine | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with omeprazole | Up to Day 63
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with ecopipam | Up to Day 63
  Subjects will be continually monitored for adverse events
Absolute values of white blood cell (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets (1000/mm3) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Absolute values of hematocrit (percent) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Absolute values of hemoglobin (g/dL) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Absolute values of Red blood cell (RBC) count (M/mm3) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Absolute values of sodium, potassium, chloride (mmol/L) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Absolute values of magnesium, urea, phosphorus, calcium, glucose, and total, conjugated and unconjugated bilirubin (mg/dL) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Absolute values of albumin and total protein (g/dL) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Absolute values of alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), creatinine phosphokinase (CPK), and creatinine (U/L) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Absolute values of urine specific gravity | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine pH | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine glucose | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine protein | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine blood | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine ketones | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine bilirubin and nitrite | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urobilinogen (Eu/dL) | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of urine leukocytes by dipstick | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge white blood cell (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets (1000/mm3) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day -1 to Day of Discharge in hematocrit (percent) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day -1 to Day of Discharge in hemoglobin (g/dL) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day -1 to Day of Discharge in Red blood cell (RBC) count (M/mm3) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day -1 to Day of Discharge in sodium, potassium, chloride (mmol/L) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Change from Day -1 to Day of Discharge in magnesium, urea, phosphorus, calcium, glucose, and total, conjugated and unconjugated bilirubin (mg/dL) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Change from Day -1 to Day of Discharge in albumin and total protein (g/dL) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Change from Day -1 to Day of Discharge in alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and creatinine phosphokinase (CPK), and creatinine (U/L) | Up to Day 26
  Blood samples will be collected for the assessment of clinical chemistry parameters
Change from Day -1 to Day of Discharge in urine specific gravity | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine pH | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine glucose | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine protein | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine blood | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine ketones | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine bilirubin and nitrite | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urobilinogen (Eu/dL) | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Change from Day -1 to Day of Discharge in urine leukocytes by dipstick | Up to Day 26
  Urine samples will be collected for the assessment of urine parameters
Absolute values of electrocardiogram (ECG) parameters: PR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) (Milliseconds) | Up to Day 26
  Twelve-lead ECGs will be obtained with the participant in a supine position after a rest of at least 5 minutes using an automated ECG machine. PR, QRS, QT, and QTcF intervals will be measured
Change from pre-dose for the respective day in ECG parameters: PR, QRS, QT, and QTcF (Milliseconds) | Up to Day 26
  Twelve-lead ECGs will be obtained with the participant in a supine position after a rest of at least 5 minutes using an automated ECG machine. PR, QRS, QT, and QTcF intervals will be measured
Absolute values of oral temperature (degrees Celsius) | Up to Day 26
  Temperature will be assessed as part of vital signs
Change from pre-dose for the respective day in oral temperature (degrees Celsius) | Up to Day 26
  Temperature will be assessed as part of vital signs
Absolute values of heart rate (beats/minute) | Up to Day 26
  Heart rate will be assessed as part of vital signs
Change from pre-dose for the respective day in heart rate (beats/minute) | Up to Day 26
  Heart rate will be assessed as part of vital signs
Absolute values of respiratory rate (breaths/minute) | Up to Day 26
  Respiratory rate will be assessed as part of vital signs
Absolute values of systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHG) | Up to Day 26
  Blood pressure will be assessed as part of vital signs
Change from pre-dose for the respective day in SBP and DBP (mmHG) | Up to Day 26
  Blood pressure will be assessed as part of vital signs
Absolute values of mean corpuscular hemoglobin (MCH) (pg) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day 1 to Day of Discharge of mean corpuscular hemoglobin (MCH) (pg) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Absolute values of mean corpuscular volume (MCV) (fL) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day 1 to Day of Discharge of mean corpuscular volume (MCV) (fL) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Absolute values of mean corpuscular hemoglobin concentration (MCHC) (g/dL) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters
Change from Day 1 to Day of Discharge of mean corpuscular hemoglobin concentration (MCHC) (g/dL) | Up to Day 26
  Blood samples will be collected for the assessment of hematology parameters

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No